CLINICAL TRIAL: NCT07218406
Title: Comparison of Merit Prelude Ideal and Terumo Glidesheath Slender Radial Artery Sheaths
Status: Not yet recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-Radial Artery Sheaths
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Transradial Access
Keywords: transradial access; randomized trial; pragmatic EMR-based trial; TRA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Terumo Glidesheath Slender sheath: Physicians will use the Terumo Glidesheath Slender sheath during the procedure.
  Interventions: Device: Terumo Glidesheath Slender sheath
- Merit Prelude Ideal sheath: Physicians will use the Merit Prelude Ideal sheath during the procedure.
  Interventions: Device: Merit Prelude Ideal sheath

INTERVENTIONS:
Device: Terumo Glidesheath Slender sheath — Terumo Glidesheath Slender sheath in the radial artery
  Groups: Terumo Glidesheath Slender sheath
Device: Merit Prelude Ideal sheath — Merit Prelude Ideal sheath in the radial artery
  Groups: Merit Prelude Ideal sheath

SUMMARY:
The aim of this study is to determine physician preference of sheath type based on a qualitative survey utilizing an EPIC-based randomization platform.

DETAILED DESCRIPTION:
Physician's with patients undergoing diagnostic coronary angiography or percutaneous coronary intervention (PCI) via a planned radial artery access approach will be randomized to either the Terumo Glidesheath Slender or Merit Prelude Ideal radial artery sheath via an electronic medical record (EMR) (EPIC)-based randomization that will be conducted automatically prior to the procedure. The nursing team will set up the room as per usual and include the sheath that was identified in the randomization process. Physician's will complete the diagnostic coronary angiography and/or PCI per usual standard of care. Physicians will complete the questionnaire regarding their preferences at the end of the case. With the exception of the physician survey, the data to be reviewed will already exist as part of the standard EMR documentation. Datacore analysts will retrieve data of patients randomized from the EMR and populate in a database for analysis using a unique identifier that does not link the patients to their identifiable information (i.e. de-identified).

ELIGIBILITY:
Inclusion Criteria:

* Physician has patient(s) undergoing diagnostic coronary angiography or percutaneous coronary intervention (PCI) across the NYU Langone Health enterprise will be eligible for the study.

Exclusion Criteria:

* No plan for at least one radial artery access
* Physician preference to not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians within the NYU Cardiac Catheterization Laboratory
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Physicians satisfaction score | Within one day of procedure
  Outcome measure is assessed by the Qualitative survey of physician satisfaction. The survey asks physicians to rate 6 items from 1 being the worst (very bad) to 5 being the best (very good) about the radial artery sheath used in their case. Total scores range from 6-30, with higher scores indicating greater satisfaction with the device.

SECONDARY OUTCOMES:
Requirement of a skin nick to advance the sheath (yes/no) | Within one day of procedure
  Outcome measure is assessed by the Qualitative survey of physician satisfaction. Binary outcome of yes or no
Presence of leakage from the sheath's hemostatic valve during the procedure (yes/no) | Within one day of procedure
  Outcome measure is assessed by the Qualitative survey of physician satisfaction. Binary outcome of yes or no based on qualitative survey
Number of cases with radial artery spasm | Within one day of procedure
  Outcome measure is assessed by the Qualitative survey of physician satisfaction.
Number of cases with patient reported forearm pain | Within one day of procedure
  Outcome measure is assessed by the Qualitative survey of physician satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Rao, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a quality improvement (QI) project under the institution's quality improvement oversight committee and individual participant data (IPD) will not be shared with other researchers.